CLINICAL TRIAL: NCT06796855
Title: Selective Bladder Denervation vs Intramuscular Onabotulinum Toxin A for Refractory Overactive Bladder: A Randomized Comparative Study
Brief Title: Comparing Treatments for Refractory Overactive Bladder: Bladder Denervation vs Botulinum Toxin Injections
Acronym: SBD-BOT-OAB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bagcilar Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Bagcilar Training and Research
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2024-12

CONDITIONS: Overactive Bladder Syndrome; Refractory Overactive Bladder
Keywords: Onabotulinum Toxin A; Selective Bladder Denervation; RF Ablation; Overactive Bladder; Intravesical Botox
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Intervention Model Description: This study uses a parallel design, where participants are randomly assigned to one of two groups for the duration of the study. The two groups are:
  The Selective Bladder Denervation group, which undergoes treatment with radiofrequency ablation (RFA).
  The Intravesical Onabotulinum Toxin A group, which receives onabotulinum toxin A injections into the bladder wall.
  Each group receives its respective intervention without crossover between treatments. Randomization was performed using the "Research Randomizer" tool to ensure an unbiased allocation of participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Selective Bladder Denervation via Radiofrequency Ablation (Experimental): Participants in this arm will undergo selective bladder denervation using a radiofrequency ablation procedure. This minimally invasive treatment involves applying controlled radiofrequency energy at four submucosal points in the bladder trigone area under general anesthesia. The procedure aims to reduce nerve overactivity and improve symptoms of refractory overactive bladder. Follow-up assessments will evaluate symptom improvement, safety, and quality of life over a 3-month period.
  Interventions: Device: Selective Bladder Denervation via Radiofrequency Ablation
- Intravesical Onabotulinum Toxin A Injection (Active Comparator): Participants in this arm will receive intravesical injections of Onabotulinum toxin A. A total of 100 units will be injected into 10 sites on the bladder wall under local anesthesia. This intervention is an established third-line treatment for refractory overactive bladder, aimed at reducing bladder overactivity. Symptom improvement, safety, and quality of life will be assessed during follow-up visits over a 3-month period.
  Interventions: Drug: Intravesical Onabotulinum Toxin A Injection

INTERVENTIONS:
Device: Selective Bladder Denervation via Radiofrequency Ablation — Participants in this arm will undergo a single session of selective bladder denervation using radiofrequency ablation (RFA). The procedure is performed under general anesthesia using the Apro Korea AK-F200 system, which delivers radiofrequency energy at four submucosal points in the bladder trigone area. The energy is applied at 25 watts per site for 60 seconds, targeting nerve pathways involved in overactive bladder symptoms. The procedure is conducted using a 19 Fr. rigid cystoscope in lithotomy position, ensuring precise electrode placement. Patients are discharged on postoperative day 1 following urinary ultrasound and post-void residual (PVR) assessment. Follow-up visits are scheduled at 2, 4, and 12 weeks to evaluate symptom improvement and safety.
  Arms: Selective Bladder Denervation via Radiofrequency Ablation
Drug: Intravesical Onabotulinum Toxin A Injection — Participants in this arm will receive a single dose of 100 units of Onabotulinum Toxin A injected into 10 sites on the bladder wall using a 4mm injection needle and 19 Fr. rigid cystoscope. The injection is administered under local anesthesia in an outpatient setting. The Onabotulinum Toxin A is diluted in sterile saline and delivered into the detrusor muscle, aiming to reduce detrusor overactivity and urgency symptoms. Patients undergo urinary ultrasound and post-void residual volume (PVR) assessment on postoperative day 1 before discharge. No additional doses are administered, and follow-up visits are scheduled at 2, 4, and 12 weeks to evaluate symptom improvement and safety.
  Arms: Intravesical Onabotulinum Toxin A Injection

SUMMARY:
The goal of this clinical trial is to compare the effectiveness and safety of two treatments for refractory overactive bladder in adult women.

The main questions it aims to answer are:

* Does selective bladder denervation using radiofrequency ablation improve overactive bladder symptoms more effectively than intravesical Onabotulinum toxin A injections?
* What are the safety profiles of each treatment?

Researchers will compare selective bladder denervation using radiofrequency ablation to intravesical Onabotulinum toxin A injections to determine which treatment is more effective and tolerable for patients whose symptoms persist despite behavioral and medical therapies.

Participants will:

* Be women aged 18 and older diagnosed with overactive bladder who did not benefit from at least two prior medical treatments for 3 months or were unable to tolerate those treatments.
* Be randomly assigned to receive either radiofrequency ablation or Onabotulinum toxin A treatment.
* Attend follow-up visits at weeks 2, 4, and 12 over a 3-month period, during which symptom improvement will be assessed using validated questionnaires and side effects will be monitored through imaging, blood, and urine tests.

DETAILED DESCRIPTION:
This randomized clinical trial aims to evaluate the effectiveness and safety of two third-line treatment options for women with refractory overactive bladder syndrome: selective bladder denervation using radiofrequency ablation and intravesical Onabotulinum toxin A injection.

The study includes 60 symptomatic female patients aged 18 years and older who met the eligibility criteria and had either failed to achieve adequate symptom control with at least two different oral pharmacological treatments or were unable to tolerate such therapies. Participants were randomly assigned into two equal groups, with 30 patients in each group, using the "Research Randomizer" tool.

Participant Assessments:

At the initial assessment, all participants underwent the following evaluations:

* A detailed medical history, including past surgeries and prior medication use.
* Urinary tests, including urinalysis and urine culture, as well as blood biochemical evaluations.
* Imaging with urinary system ultrasonography to evaluate both the upper and lower urinary tract and measure post-void residual urine volume.
* Symptom assessment using the following validated patient-reported outcome questionnaires:

International Consultation on Incontinence Questionnaire - Female Lower Urinary Tract Symptoms (ICIQ-FLUTS).

Overactive Bladder Symptom Score Questionnaire (OAB-V8). Incontinence Quality of Life Questionnaire (I-QOL).

Additionally, participants were asked to maintain a three-day bladder diary to document:

* The number of daily urinations.
* Episodes of waking up at night to urinate (nocturia).
* Urgency episodes.
* Instances of urge urinary incontinence.

Treatment Groups:

1. Selective Bladder Denervation with Radiofrequency Ablation:

   This procedure was performed under general anesthesia using the Apro Korea AK-F200 radiofrequency system, which operates with temperature and impedance control along with a cooling mechanism.

   Radiofrequency energy was applied to four specific submucosal points in the bladder's trigone region.

   The target tissue temperature was 100 degrees Celsius, with energy delivery set to 25 watts for 60 seconds at each point.

   Post-procedure imaging and post-void residual urine measurements were performed to ensure patient safety.
2. Intravesical Onabotulinum Toxin A Injection:

This treatment was administered under local anesthesia using a rigid cystoscope.

A total dose of 100 units of Onabotulinum toxin A was injected into ten separate points across the bladder wall.

Follow-Up Protocol:

Patients were scheduled for follow-up visits at 2, 4, and 12 weeks after the intervention. At each visit, the following evaluations were conducted:

* Ultrasonographic imaging of the urinary system to assess for any upper tract dilation (hydronephrosis) and to measure post-void residual urine volume.
* Laboratory assessments, including urinalysis and serum creatinine level evaluation.
* Reassessment of urinary symptoms through a repeat three-day bladder diary and completion of the same validated patient-reported outcome questionnaires.

Study Objective:

This clinical trial aims to compare the two treatment modalities concerning their effectiveness in relieving symptoms of overactive bladder, improving patients' quality of life, and assessing their safety profiles. The results of this study are expected to provide valuable insights into the optimal third-line treatment approach for patients with refractory overactive bladder who have not responded to conventional behavioral and pharmacological therapies.

ELIGIBILITY:
Inclusion Criteria:

Biological females aged 18 years or older.

Diagnosis of refractory overactive bladder syndrome, defined as:

* Persistent symptoms despite having completed behavioral therapy and at least two different oral pharmacotherapies (e.g., anticholinergics or beta-3 adrenergic agonists) for a minimum of 3 months each; or
* Inability to tolerate oral pharmacotherapy for overactive bladder syndrome. Willingness and ability to provide written informed consent. Ability to comply with the study protocol, including attendance at scheduled follow-up visits and completion of validated symptom assessment questionnaires (e.g., Overactive Bladder Symptom Score - OAB-V8, International Consultation on Incontinence Questionnaire - Female Lower Urinary Tract Symptoms - ICIQ-FLUTS).

Exclusion Criteria:

Pregnancy or intention to become pregnant within 12 months of enrollment. History of stress urinary incontinence as the predominant symptom.

Recent interventions prior to enrollment:

* Oral medication for overactive bladder within the past 2 weeks.
* Intravesical Onabotulinum toxin A injection within the past 9 months.
* Pelvic electrical stimulation within the past 2 weeks. Active or chronic urinary tract infection or a history of urinary retention within the past 6 months.

Active hematuria or known bleeding disorders.

History or current diagnosis of:

* Bladder cancer or ongoing bladder cancer treatment.
* Bladder outlet obstruction, ureteral dysfunction, ureteral stricture, or vesicoureteral reflux.
* Elevated serum creatinine level (≥2 times the upper limit of normal) within the past 6 months.

Neurological conditions affecting bladder function, including but not limited to:

* Multiple sclerosis.
* Myasthenia gravis.
* Spinal cord injury or disease. Any condition deemed by the investigator to interfere with study participation or accurate evaluation of outcomes.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Overactive Bladder Assessment Tool (OAB-V8) Total Score at 12 Weeks | From baseline to 12 weeks post-treatment
  The Overactive Bladder Assessment Tool (OAB-V8) is an 8-item validated questionnaire used to assess the severity of overactive bladder (OAB) symptoms, including urinary urgency, frequency, nocturia, and urge urinary incontinence.
  Each item is rated on a 6-point Likert scale from 0 (not at all) to 5 (a very severe problem), resulting in a total score ranging from 0 to 40, with higher scores indicating greater symptom severity.
  The primary outcome of this study is the change from baseline in OAB-V8 total score at 12 weeks. A clinically significant response is defined as a ≥50% reduction in total OAB-V8 score compared to baseline.

SECONDARY OUTCOMES:
Change from Baseline in International Consultation on Incontinence Questionnaire - Female Lower Urinary Tract Symptoms (ICQ-FLUTS) Score at 12 Weeks | From baseline to 12 weeks post-treatment
  The International Consultation on Incontinence Questionnaire - Female Lower Urinary Tract Symptoms (ICIQ-FLUTS) is a validated tool used to assess lower urinary tract symptoms and their impact on quality of life in female patients. It consists of three domains:
  Filling symptoms (e.g., urgency, frequency) Voiding symptoms (e.g., hesitancy, weak stream) Incontinence symptoms (e.g., stress or urgency incontinence)
  Each item is scored on a 4-point Likert scale (0 to 3), with higher scores indicating greater symptom severity. The total score ranges from 0 to 48.
  The secondary outcome is the change in ICIQ-FLUTS total score from baseline to 12 weeks. Improvement is defined as a reduction of 30% or more in the total score.
Change from Baseline in Incontinence Quality of Life (I-QOL) Score at 12 Weeks | From baseline to 12 weeks post-treatment
  The Incontinence Quality of Life (I-QOL) questionnaire is a 26-item validated tool assessing the impact of urinary incontinence on daily activities, emotional well-being, and social interactions.
  Each item is rated on a 5-point Likert scale (1 = extremely, 5 = not at all). The total score ranges from 0 to 100, with higher scores indicating better quality of life.
  The secondary outcome is the change in I-QOL score from baseline to 12 weeks. A clinically significant improvement is defined as an increase of 10 points or more.
Change from Baseline in Urgency and Urgency Urinary Incontinence (UUI) Episodes at 12 Weeks | From baseline to 12 weeks post-treatment
  The number of urgency episodes and urgency incontinence episodes per 24-hour period will be recorded using a patient-reported bladder diary.
  A clinically significant improvement is defined as a ≥50% reduction in urgency or urge urinary incontinence episodes from baseline.
Incidence of Treatment-Related Adverse Events at 12 Weeks | From baseline to 12 weeks post-treatment
  The incidence and severity of treatment-related adverse events (AEs) will be documented at each follow-up visit. AEs will be classified according to Common Terminology Criteria for Adverse Events (CTCAE v5.0) and may include:
  Urinary retention Hematuria (gross or microscopic) Dysuria or pain during urination Pelvic pain or discomfort Hydronephrosis

OTHER OUTCOMES:
Change from Baseline in Daily Voiding Frequency and Nocturia Episodes at 12 Weeks | From baseline to 12 weeks post-treatment
  The total number of voiding episodes per 24 hours, including daytime and nighttime frequency (nocturia), will be assessed using a bladder diary.
  A clinically significant reduction is defined as a ≥30% decrease in daily voiding frequency and a ≥1 episode reduction in nocturia per night.
Change from Baseline in Post-Void Residual (PVR) Urine Volume at 12 Weeks | From baseline to 12 weeks post-treatment
  Post-void residual (PVR) volume will be measured using ultrasound assessment at each follow-up visit. Post-void residual is the amount of urine remaining in the bladder after voluntary voiding and is an important indicator of voiding efficiency and urinary retention risk.
  A PVR >100 mL is considered clinically significant urinary retention. The secondary outcome is the change in PVR from baseline to 12 weeks, with an increase >50 mL considered a potential adverse effect.
Incidence of Culture-Proven Urinary Tract Infections (UTIs) at 12 Weeks | From baseline to 12 weeks post-treatment
  The number of participants diagnosed with urinary tract infections will be recorded during the follow-up period.
  A symptomatic urinary tract infection is defined as the presence of a positive urine culture (≥100,000 colony-forming units per milliliter [CFU/mL]) accompanied by at least one urinary symptom, such as dysuria (painful urination), urinary frequency, urgency, or fever.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammet M Dinçer, MD, Study Director — University of Health Sciences, Istanbul Bagcilar Hospital
Locations (1):
- University of Health Sciences, Istanbul Bagcilar Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Baseline demographic data. Outcome measures (e.g., Overactive Bladder Symptom Score (OAB-V8), International Consultation on Incontinence Questionnaire - Female Lower Urinary Tract Symptoms (ICQ-FLUTS), Incontinence Quality of Life Scale (I-QOL), and Post-Void Residual (PVR) urine volume values).
  Adverse event data.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: January 2025 - January 2026
Access Criteria: Researchers from academic institutions, non-profit organizations, or industry with a valid scientific interest in the study outcomes will be eligible to access the data.
  Data will be shared with researchers upon request, subject to:
  * Submission of a written proposal outlining the research objectives.
  * Review and approval by the study investigators.
  Interested researchers can contact the principal investigator at:
  Email: zekisonmez91@gmail.com Phone: +90 505 6101066

REFERENCES:
- [Background] Rovner ES, Versi E, Le Mai T, Dmochowski RR, De Wachter S. One-year results with selective bladder denervation in women with refractory overactive bladder. Neurourol Urodyn. 2019 Nov;38(8):2178-2184. doi: 10.1002/nau.24110. Epub 2019 Jul 29. PMID 31359508
- [Background] Fugett J 2nd, Phillips L, Tobin E, Whitbrook E, Bennett H, Shrout J, Coad JE. Selective bladder denervation for overactive bladder (OAB) syndrome: From concept to healing outcomes using the ovine model. Neurourol Urodyn. 2018 Sep;37(7):2097-2105. doi: 10.1002/nau.23560. Epub 2018 Mar 31. PMID 29603776
- [Background] Tu LM, De Wachter S, Robert M, Dmochowski RR, Miller LE, Everaert K. Initial clinical experience with selective bladder denervation for refractory overactive bladder. Neurourol Urodyn. 2019 Feb;38(2):644-652. doi: 10.1002/nau.23881. Epub 2018 Nov 29. PMID 30499155